CLINICAL TRIAL: NCT02985645
Title: Graftless Maxillary Sinus Augmentation With CGF Utilizing DIVA System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, ruth angel dar, Principal Investigator, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0153-16-NHR
Record Dates: First submitted 2016-11-26; First posted 2016-12-07 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Alveolar Bone Loss
Keywords: CGF; sinus augmentation; DIVA; Platelet-Rich Plasma
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): maxillary sinus augmentation with CGF
  Interventions: Procedure: maxillary sinus augmentation with CGF; Device: "dynamic implant valve approach" - DIVA system

INTERVENTIONS:
Procedure: maxillary sinus augmentation with CGF — Graftless maxillary sinus augmentation surgery with CGF application utilizing DIVA system
Device: "dynamic implant valve approach" - DIVA system — The DIVA system will be used to apply the CGF to the maxillary sinus.

SUMMARY:
This study is intended to evaluate the efficiency of graftless maxillary sinus augmentation with concentrated growth factor (CGF) utilizing "dynamic implant valve approach" (DIVA) system.

DETAILED DESCRIPTION:
Crestal bone deficiency in the posterior maxilla may present a therapeutic challenge when dental implants are required. Sufficient bone volume is necessary for the long term survival of the implant .

The two most used surgical techniques are the crestal and the lateral window. The latter was first described by Tatum and subsequently, Boyene and James in 1980 . In the original technique, after fracturing the sinus floor, an implant was placed and submerged during the healing phase. The crestal osteotome technique is less invasive and was first described by Summers in 1994 . In this technique, a set of osteotomes is used to prepare the implant site, thereby allowing bone preservation.

Since the sinus augmentation was describes, bone grafts have been the mainstay of treatment. Variable bone grafts, such as autografts, allografts, xenografts, alloplasts, or combinations of different graft materials, have been used widely with similar results . Nonetheless, successful bone augmentation in the maxillary sinus, without bone grafting, have been reported in human and animal studies.

In 2011, Dong-Seok et al described sinus augmentation through a lateral window approach, using a fibrin rich block with concentrated growth factor (CGF). The researchers showed successful new bone formation in the sinus, with a success rate of 98% and no major complications .

Graftless Sinus augmentation relies on bioactive mediators that stimulate cell proliferation, matrix remodeling, and angiogenesis. CGF is one of the latest developments in this field, and is produced by processing blood samples with a special centrifuge device. It contains several mediators - platelet-derived growth factor (PDGF), transforming growth factor-b1 (TGF-b1) and b2 (TGF-b2), fibroblast growth factor (FGF), vascular endothelial growth factor (VEGF), and insulin-like growth factor (IGF). Because CGF is a dense fibrin matrix, richer in growth factors than other preparations, it has proved to have a better regenerative capacity and versatility .

As for the application of CGF, the introduction of the "dynamic implant valve approach" (DIVA), a minimally invasive approach procedure, enables the use of a closed bone augmentation technique. The implant was designed with an internal sealing screw that might serve as drug delivery system via its channel.

In this study, a graftless maxillary sinus augmentation with CGF will be performed utilizing DIVA system, and the bone formation will be periodically measured using panoramic X-ray and cone beam computerized tomography (CBCT).

In addition, in vitro cumulative release of selected growth factors of the CGF will be analyzed. The total quantity of growth factors will be checked using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* No medical history of diseases involving bone metabolism
* Patients that are treated by a prostodontist
* Healthy oral cavity and sinuses, and good oral hygiene
* No bone pathology demonstrated by X-ray
* Residual sub-antral bone of at least 4mm as demonstrated by computerized tomography (CT)
* The patient does not participate in another clinical study
* The patient can read and understand the informed consent

Exclusion Criteria:

* Medical history of a disease affecting bone metabolism (Diabetes Mellitus, heart disease, renal failure, osteoporosis)
* Medical treatment that can affect bone metabolism (such as Bisphosphonates)
* Patients treated with anticoagulants (such as Coumadin, Pradaxa)
* Personal history of chemotherapy or radiotherapy
* Patients with maxillary sinus pathology
* Patients lacking a prostodontic treatment plan
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
bone formation after sinus augmentation | one year
  during postoperative follow-up, bone formation in the maxillary sinus will be assessed by periodic imaging.
  after one year the investigators expect to see complete implant integration into the bone formed in the maxillary sinus(e.g; the dental implant is completely covered by bone).

SECONDARY OUTCOMES:
Quantification of growth factors released from the CGF matrix in vitro | one year
  ELISA test will be used to quantify the released growth factors, and the data will be compared to the factors released from regular bone material.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Srouji, Prof., Study Director — Western Galilee Medical Center
Locations (1):
- Western Galilee Medical Center, Nahariya, Israel

REFERENCES:
- [Background] Del Fabbro M, Corbella S, Weinstein T, Ceresoli V, Taschieri S. Implant survival rates after osteotome-mediated maxillary sinus augmentation: a systematic review. Clin Implant Dent Relat Res. 2012 May;14 Suppl 1:e159-68. doi: 10.1111/j.1708-8208.2011.00399.x. Epub 2011 Nov 14. PMID 22082056
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Summers RB. The osteotome technique: Part 3--Less invasive methods of elevating the sinus floor. Compendium. 1994 Jun;15(6):698, 700, 702-4 passim; quiz 710. PMID 7994726
- [Background] Danesh-Sani SA, Loomer PM, Wallace SS. A comprehensive clinical review of maxillary sinus floor elevation: anatomy, techniques, biomaterials and complications. Br J Oral Maxillofac Surg. 2016 Sep;54(7):724-30. doi: 10.1016/j.bjoms.2016.05.008. Epub 2016 May 25. PMID 27235382
- [Background] Falah M, Sohn DS, Srouji S. Graftless sinus augmentation with simultaneous dental implant placement: clinical results and biological perspectives. Int J Oral Maxillofac Surg. 2016 Sep;45(9):1147-53. doi: 10.1016/j.ijom.2016.05.006. Epub 2016 May 31. PMID 27256011
- [Background] Sohn DS, Kim WS, An KM, Song KJ, Lee JM, Mun YS. Comparative histomorphometric analysis of maxillary sinus augmentation with and without bone grafting in rabbit. Implant Dent. 2010 Jun;19(3):259-70. doi: 10.1097/ID.0b013e3181df1406. PMID 20523182
- [Background] Sohn DS, Heo JU, Kwak DH, Kim DE, Kim JM, Moon JW, Lee JH, Park IS. Bone regeneration in the maxillary sinus using an autologous fibrin-rich block with concentrated growth factors alone. Implant Dent. 2011 Oct;20(5):389-95. doi: 10.1097/ID.0b013e31822f7a70. PMID 21881519
- [Background] Rodella LF, Favero G, Boninsegna R, Buffoli B, Labanca M, Scari G, Sacco L, Batani T, Rezzani R. Growth factors, CD34 positive cells, and fibrin network analysis in concentrated growth factors fraction. Microsc Res Tech. 2011 Aug;74(8):772-7. doi: 10.1002/jemt.20968. PMID 21780251
- [Background] Nahlieli O. Dynamic implant valve approach for dental implant procedures. Chin J Dent Res. 2014;17(1):15-21. PMID 25028685